CLINICAL TRIAL: NCT02843009
Title: Overcoming the Blunted Response to Resistance Exercise With Fish Oil to Maximise Musculoskeletal Properties and Functional Abilities in Older People
Brief Title: Fish Oil and Adaptations to Resistance Exercise in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Dr, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gray BBSRC NI
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Ageing
MeSH Terms: interventions — Resistance Training; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safflower Oil plus Resistance Exercise Training (Placebo Comparator): 3.0g of safflower oil taken daily alongside twice weekly resistance exercise training sessions for 18 weeks
  Interventions: Behavioral: Resistance Exercise Training; Dietary Supplement: Supplementation
- Fish Oil plus Resistance Exercise Training (Active Comparator): 3.0g of fish oil taken daily alongside twice weekly resistance exercise training sessions for 18 weeks
  Interventions: Behavioral: Resistance Exercise Training; Dietary Supplement: Supplementation

INTERVENTIONS:
Behavioral: Resistance Exercise Training — Resistance exercise will involve 2 sessions per week for 18 weeks. Each session will involve participants carrying out the following exercises: calf press, leg press, leg extension and leg curl
Dietary Supplement: Supplementation — Participants randomised to either 3g/day of fish oil or safflower oil for 18 weeks

SUMMARY:
Skeletal muscle is the largest organ in the human body and has many important roles in determining our physical abilities and overall wellbeing. One major function of skeletal muscle is to carry out many daily tasks, such as rising from a chair or getting on a bus, tasks often referred to as functional abilities. During healthy ageing muscle size is reduced by approximately 0.5-2% a year (known as sarcopenia), with concurrent reductions in functional abilities. This can result in a reduction in quality of life and loss of independence, both of which are clearly not desirable. The incidence of sarcopenia is around 20% between 50-70 years and around 50% in those over 80 years, with the absolute numbers and the average age of the population rising. One method through which muscle function can be enhanced and retard the progression of sarcopenia, across all age groups, is through exercise. The effectiveness of exercise will depend on a number of genetic and environmental factors, with nutritional intake being one of the most important and easily altered. Recent research has suggested that altering the type of fatty acids consumed may have a positive effect on muscle function. Little research is yet to be carried out in elderly humans. This is important as that findings from animal models are not definitively transferrable to humans. The main aim of the current proposal, therefore, is to investigate the effect the consumption of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), long chain polyunsaturated fatty acids found in oily fish, on the response to a resistance training programme in the elderly. A further aim is to determine the mechanisms which result in these adaptive responses. The project will be centred round a large 18 week resistance training/nutritional (EPA/DHA) intervention with both males and females over the age of 65 years. There are three main research questions and experiments stemming from this intervention. 1) Does the consumption of EPA and DHA result in a greater increase in strength, power and functional abilities in response to resistance training? To answer this question a series of measures of muscular performance and functional abilities will be assessed. 2) Does the consumption of EPA and DHA increase the size and quality of muscles, reduce the amount of fat found within the muscle and decrease inflammation? To address this question the participants will have MRI images of their muscles and blood samples taken before and after the intervention. This will allow the calculation of muscle mass/fat content and circulating levels of inflammatory markers. 3) Does the consumption of EPA and DHA enhance the activity of the molecules involved in controlling muscle mass after a single bout of resistance exercise? For this question muscle samples will be obtained before and after a single training session and measure changes in molecules previously identified as important in the changes in muscle mass in response to exercise. A fourth aim running throughout the proposal is 4) Do males and females respond differently to the combination of EPA/DHA and resistance exercise? Differences in protein metabolism have previously been noted between genders and yet the investigation of these differences is often overlooked. The investigators will investigate this by studying responses in groups of males and females. In summary, the aim of the proposed project is to test the hypothesis that the consumption of fatty acids found in oily fish will improve the response of an elderly population to a resistance training intervention. The major outcome of the proposal would be in establishing a beneficial effect of fish oil on muscular adaptation in the elderly, opening up a widely available therapeutic strategy for an improvement in the quality of life in the elderly population. Such strategies are of particular importance due to the increasing age of the UK population.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years of age
* Not consuming oily fish regularly
* Not consuming nutritional supplements
* Not participating in resistance exercise training

Exclusion Criteria:

* History of myocardial infarction within previous 2 years
* Cardiac illness: moderate/ severe aortic stenosis, acute pericarditis, acute myocarditis, aneurysm, severe angina, clinically significant valvular disease, uncontrolled dysrhythmia, claudication within the previous 10 years
* Thrombophlebitis or pulmonary embolus within the previous 2 years
* History of cerebrovascular disease (CVA or TIA) within the previous 2 years
* Acute febrile illness within the previous 3 months
* Severe airflow obstruction
* Uncontrolled metabolic disease (e.g., thyroid disease or cancer)
* Significant emotional distress, psychotic illness or depression within the previous 2 years
* Lower limb fracture sustained within the previous 2 years; upper limb fracture within the previous 6 months; non arthroscopic lower limb joint surgery within the previous 2 years
* Any reason for loss of mobility for greater than 1 week in the previous 2 months or greater than 2 weeks in the previous 6 months
* Poorly controlled atrial fibrillation
* Poor (chronic) pain control
* Resting systolic pressure >200 mmHg or resting diastolic pressure >100 mmHg
* Moderate/ severe cognitive impairment (MMSE <23)
* Impaired tissue viability (defined by a Waterlow risk assessment score >15).

Based on Greig C.A. et al. Age Ageing 1994, 23: 185-9

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximal Isometric Knee Extensor Torque | Change from baseline at 18 weeks

SECONDARY OUTCOMES:
Short Performance Physical Battery Test | Change from baseline at 18 weeks
Maximal Isokinetic Knee Extensor Torque (30,90 and 120 degrees/s) | Change from baseline at 18 weeks
Quadriceps Cross Sectional Area (MRI) | Change from baseline at 18 weeks
Circulating markers of inflammation (IL-6 and TNF-alpha) | Change from baseline at 18 weeks
Muscle protein synthesis | 18 weeks
Muscle P70s6k activity | Change from baseline to 2h post-exercise
Erythrocyte fatty acid composition | Change from baseline at 18 weeks
Muscle membrane fatty acid composition | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Da Boit M, Tommasi S, Elliot D, Zinellu A, Sotgia S, Sibson R, Meakin JR, Aspden RM, Carru C, Mangoni AA, Gray SR. Sex Differences in the Associations between L-Arginine Pathway Metabolites, Skeletal Muscle Mass and Function, and their Responses to Resistance Exercise, in Old Age. J Nutr Health Aging. 2018;22(4):534-540. doi: 10.1007/s12603-017-0964-6. PMID 29582894
- [Derived] Da Boit M, Sibson R, Sivasubramaniam S, Meakin JR, Greig CA, Aspden RM, Thies F, Jeromson S, Hamilton DL, Speakman JR, Hambly C, Mangoni AA, Preston T, Gray SR. Sex differences in the effect of fish-oil supplementation on the adaptive response to resistance exercise training in older people: a randomized controlled trial. Am J Clin Nutr. 2017 Jan;105(1):151-158. doi: 10.3945/ajcn.116.140780. Epub 2016 Nov 16. PMID 27852617